CLINICAL TRIAL: NCT00985517
Title: A Phase 1/2 Trial Assessing the Safety and Efficacy of Bilateral Intraputaminal and Intranigral Administration of CERE-120 (Adeno-Associated Virus Serotype 2 [AAV2]-Neurturin [NTN]) in Subjects With Idiopathic Parkinson's Disease
Brief Title: Safety and Efficacy of CERE-120 in Subjects With Parkinson's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sangamo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CERE-120-09
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Results first posted 2020-03-26 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Parkinson's disease; Movement Disorders; Gene Therapy; Neurotrophic Factors; GDNF; Neurturin; DBS; Dopamine
MeSH Terms: conditions — Parkinson Disease; Movement Disorders

STUDY DESIGN:
Intervention Model Description: In the first part of the study (Phase 1), 2 escalating dose cohorts received CERE-120.
  In the second part of the study (Phase 2), subjects were randomized 1:1 to receive CERE-120 or Sham Surgery.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phase 1: Cohort 1 (Experimental): CERE-120 9.4 x 10^11 vg, injected by a neurosurgeon directly in the substantia nigra and in the putamen
  Interventions: Biological: CERE-120: Adeno-Associated Virus Delivery of Neurturin
- Phase 1: Cohort 2 (Experimental): CERE-120 2.4 x 10^12 vg, injected by a neurosurgeon directly in the substantia nigra and in the putamen
  Interventions: Biological: CERE-120: Adeno-Associated Virus Delivery of Neurturin
- Phase 2: CERE-120 (Experimental): CERE-120 2.4 x 10^12 vg, injected by a neurosurgeon directly in the substantia nigra and in the putamen
  Interventions: Biological: CERE-120: Adeno-Associated Virus Delivery of Neurturin
- Phase 2: Sham Surgery (Sham Comparator): Neurosurgical procedure that mimics the procedure for CERE-120 delivery. No injections were administered during sham surgery.
  Interventions: Procedure: Sham Surgery

INTERVENTIONS:
Biological: CERE-120: Adeno-Associated Virus Delivery of Neurturin
  Other Names: AAV2-Neurturin
  Arms: Phase 1: Cohort 1; Phase 1: Cohort 2; Phase 2: CERE-120
Procedure: Sham Surgery
  Arms: Phase 2: Sham Surgery

SUMMARY:
The purpose of this study was to evaluate the safety and potential benefits of CERE-120 in the treatment of Parkinson's disease.

DETAILED DESCRIPTION:
CERE-120 is an experimental drug that consists of an adeno-associated virus (AAV) that was engineered to carry the human gene for neurturin, a neurotrophic (growth) factor. Similar to other growth factors (such as GDNF), neurturin is capable of restoring function and protecting brain cells from further damage. The virus used in CERE-120 is not known to cause disease in people.

CERE-120 is delivered directly to the brain cells most affected in Parkinson's disease - the dopamine producing neurons. CERE-120 is injected during brain surgery. Once in place, CERE-120 continuously produces neurturin.

During the first, open-label, part of the study (Phase 1), subjects with Parkinson's disease received CERE-120 at one of two dose levels. In the second part of the study (Phase 2), subjects were randomized 1:1 to receive CERE-120 or a "sham" surgery where no medication was injected.

Participants in both phases of the study were followed for up to five years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ages 35 to 70 years old (inclusive)
* A diagnosis of idiopathic Parkinson's disease based on UK Brain Bank criteria, including bradykinesia and at least 1 of the following PD features: resting tremor or rigidity
* A Hoehn and Yahr score of no greater than 3 in the "off" condition at Screening
* A robust response to dopaminergic therapy as judged by the investigator based on the UPDRS Part III: Motor Examination
* Experiencing motor complications despite adequate antiparkinsonian therapy
* A stable, optimized regimen of antiparkinsonian medications and stable parkinsonian features for at least 6 weeks prior to Screening
* Subject is willing not to undergo DBS for at least 12 months after the study surgical procedure (Phase 1 subjects) or while the study is blinded (Phase 2 subjects) and the investigator believes that this is medically acceptable
* Medically fit to undergo the study surgical procedure as determined by medical history, clinical and laboratory evaluations, and any other pre-surgical evaluations that are standard at the institution where the subject will undergo surgery
* Physically and mentally capable of performing all protocol-specified assessments and complying with the study visit schedule
* Subjects must be able to travel to study visits alone or able to identify a partner or caregiver who agrees to accompany the subject to the study visits
* Females of childbearing potential must have a negative β-HCG pregnancy test at Screening and again before surgery on Day 0
* All subjects, both male and female, must agree to practice adequate barrier method contraception for at least 6 months after the surgical procedure
* Provides written informed consent to participate before any study-specific procedures are conducted

Exclusion Criteria:

* Atypical or secondary parkinsonism, including, but not limited to, multiple system atrophy (MSA) or progressive supranuclear palsy
* Any subject for whom participation in the study would pose a substantial safety risk
* Any condition that would compromise the ability of the subject to undergo study procedures, including allergy to gadolinium
* Presence of any known brain abnormality that could interfere with the assessment of safety or efficacy or represents a surgical risk to the subject
* Evidence of significant brain atrophy on the Baseline MRI
* History of any cancer other than basal or squamous cell skin cancer within the 3 years prior to Screening
* Any chemotherapy, cytotoxic therapy, or immunotherapy (e.g., IL-2, IL-12, interferon) within the 3 months prior to Screening
* Any prior treatment for PD with a procedure involving intracranial surgery or implantation of a device (e.g. DBS, pallidotomy)
* Any prior treatment for a neurological or psychiatric disorders with a procedure involving the implantation of a device (e.g. spinal cord stimulator, vagus nerve stimulator)
* History of any prior gene transfer therapy
* Treatment with any investigational agent within the 3 months prior to Screening
* Anticipated need for antiplatelet agents or anticoagulation therapy, including gingko biloba, during the 10 days prior to the projected surgery date
* Any vaccinations within the 30 days prior to the projected surgery date Note: Vaccinations are not allowed for 30 days after the surgical procedure, unless deemed necessary by the investigator for the subject's well-being
* Not likely to be available for the duration of the trial, likely to be noncompliant with the protocol, or who are deemed unsuitable by the investigator for any other reason
* Participation in a previous surgical treatment study for Parkinson's disease

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2009-10-29 (Actual); Primary Completion 2014-11-09 (Actual); Study Completion 2017-11-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford School of Medicine, Palo Alto, California
  - University of California, San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Beth Israel Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Duke University, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Derived] Bartus RT, Baumann TL, Siffert J, Herzog CD, Alterman R, Boulis N, Turner DA, Stacy M, Lang AE, Lozano AM, Olanow CW. Safety/feasibility of targeting the substantia nigra with AAV2-neurturin in Parkinson patients. Neurology. 2013 Apr 30;80(18):1698-701. doi: 10.1212/WNL.0b013e3182904faa. Epub 2013 Apr 10. PMID 23576625

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Cohort 1: CERE-120 at 9.4 x 10^11 vg, injected by a neurosurgeon directly in the substantia nigra and in the putamen
- Phase 1: Cohort 2; Phase 2: CERE-120 Treatment Group: CERE-120 at 2.4 x 10^12 vg, injected by a neurosurgeon directly in the substantia nigra and in the putamen
- Phase 2: Sham Surgery: Neurosurgical procedure that mimics the procedure for CERE-120 delivery. No injections are performed during sham surgery.
Period: Overall Study
Arm/Group | Phase 1: Cohort 1 | Phase 1: Cohort 2 | Phase 2: CERE-120 Treatment Group | Phase 2: Sham Surgery
Started | 3 | 3 | 24 | 27
Completed | 3 | 3 | 23 | 24
Not Completed | 0 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Phase 2: CERE-120: CERE-120 at 2.4 x 10^12 vg, injected by a neurosurgeon directly in the substantia nigra and in the putamen
- Total: Total of all reporting groups
Arm/Group | Phase 1: Cohort 1 | Phase 1: Cohort 2 | Phase 2: CERE-120 | Phase 2: Sham Surgery | Total
Number analyzed (Participants) | 3 | 3 | 24 | 27 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 20 | 23 | 49
  >=65 years | 0 | 0 | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (3.0) | 55.4 (6.7) | 58.2 (7.0) | 58.0 (7.0) | 57.4 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 8 | 9 | 19
  Male | 3 | 1 | 16 | 18 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 2
  White | 3 | 2 | 23 | 27 | 55
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 24 | 27 | 57

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received CERE-120 Treatment
Description: Number of Participants who received CERE-120 Treatment
Time Frame: 5 years
Population: Phase 1: Cohort 1, Phase 1: Cohort 2, Phase 2: CERE-120, Phase 2: Sham Surgery
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: Cohort 2: CERE-120 at 2.4 x 10^12, injected by a neurosurgeon directly in the substantia nigra and in the putamen
Arm/Group | Phase 1: Cohort 1 | Phase 1: Cohort 2 | Phase 2: CERE-120 | Phase 2: Sham Surgery
Number analyzed (Participants) | 3 | 3 | 24 | 27
Participants | 3 | 3 | 24 | 27

2. Primary Outcome: Phase 1 and Phase 2: Change From Baseline in Motor Examination Part III Total Score in the "Off" Condition for the CERE-120 Group as Compared to the Sham Surgery Control Group at the Last Double-blind Assessment.
Description: UPDRS is a tool to evaluate the impact of symptomatic and potential disease modifying treatments. Part III focuses on 14 motor functions, assessing each on a scale from 0 (normal) to 4 (severe) with total score 0 - 56. The 5 Feb 2003 version of the UPDRS Rating was used in this trial. The total score is the sum of 14 motor functions. Change from baseline in total score is reported.
  The last double blind assessment for each subject is defined as the most recent assessment at the time when the final randomized subject completes the Month 15 Visit. The length of the double-blind follow-up period for each subject ranged from 15 to 24 months, depending on the enrollment rate.
Time Frame: Baseline, Months 15, 18, 21 and 24
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Phase 1: Cohort 1 | Phase 1: Cohort 2 | Phase 2: CERE-120 | Phase 2: Sham Surgery
Number analyzed (Participants) | 3 | 3 | 24 | 27
score on a scale
  MONTH 15 | NA [NA to NA] — Not a protocol specified timepoint | NA [NA to NA] — Not a protocol specified timepoint | -5.04 [-26.00 to 12.00] | -5.09 [-26.00 to 13.00]
  MONTH 18 | -3.67 [-5.00 to -2.00] | -7.33 [-9.00 to -4.00] | -5.21 [-29.00 to 14.00] | -3.78 [-24.00 to 15.00]
  MONTH 21 | NA [NA to NA] — Not a protocol specified timepoint | NA [NA to NA] — Not a protocol specified timepoint | -2.29 [-20.00 to 14.00] | -6.25 [-18.00 to 2.00]
  MONTH 24 | -7.00 [-18.00 to 1.00] | -4.00 [-16.00 to 10.00] | -8.80 [-28.00 to 7.00] | -5.46 [-30.00 to 13.00]

ADVERSE EVENTS:
Time Frame: 5 years after surgery
Groups:
- Phase 2: Sham Surgery Control Group: Neurosurgical procedure that mimics the procedure for CERE-120 delivery. No injuections are performed during sham surgery.
Arm/Group | Phase 1: Cohort 1 | Phase 1: Cohort 2 | Phase 2: CERE-120 Treatment Group | Phase 2: Sham Surgery Control Group
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 2/24 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 7/24 | 7/27
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 24/24 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Cohort 1 (N=3) | Phase 1: Cohort 2 (N=3) | Phase 2: CERE-120 Treatment Group (N=24) | Phase 2: Sham Surgery Control Group (N=27)
Left-sided acoustic neuroma (Nervous system disorders) | 0 | 0 | 1 (1) | 0 (0)
Worsened Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 1 (1) | 0 (0)
Symptomatic Bradycardia (Cardiac disorders) | 0 | 0 | 1 (1) | 0 (0)
Coronary Artery Stenosis, Symptomatic (Cardiac disorders) | 0 | 0 | 1 (1) | 0 (0)
Chest Pain with Activity (General disorders) | 0 | 0 | 0 (0) | 1 (1)
Generalized Weakness (General disorders) | 0 | 0 | 0 (0) | 1 (1)
Post Surgical Infection of R Great Toe (Infections and infestations) | 0 | 0 | 0 (0) | 1 (1)
Closed Head Injury Related to Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 (0) | 1 (1)
Severe Right Knee Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 (0) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 (0) | 1 (1)
Right Frontal Hemorrhage (Nervous system disorders) | 0 | 0 | 1 (1) | 0 (0)
Intracranial Hemorrhage (Nervous system disorders) | 0 | 0 | 1 (1) | 0 (0)
Acute Ischemic Stroke (Nervous system disorders) | 0 | 0 | 1 (1) | 0 (0)
Increased Parkinson's Disease Symptoms (Nervous system disorders) | 0 | 0 | 0 (0) | 1 (1)
Subdural and Subarachnoid Hemorrhage Secondary to Syncope and Motor Vehicle Accident (Nervous system disorders) | 0 | 0 | 0 (0) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 0 (0) | 1 (1)
R Great Toe Joint Fusion with Bone Graft Surgery (Surgical and medical procedures) | 0 | 0 | 0 (0) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Cohort 1 (N=3) | Phase 1: Cohort 2 (N=3) | Phase 2: CERE-120 Treatment Group (N=24) | Phase 2: Sham Surgery Control Group (N=27)
Angina Pectoris (Cardiac disorders) | 0 | 0 | 2 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary Artery Stenosis (Cardiac disorders) | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 2
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 2
Eye Swelling (Eye disorders) | 0 | 0 | 0 | 3
Eyelid Ptosis (Eye disorders) | 0 | 0 | 1 | 1
Macular Hole (Eye disorders) | 0 | 0 | 0 | 1
Pupils Unequal (Eye disorders) | 0 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 4 | 3
Dental Caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gingival Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hypoaesthesia Oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mouth Ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 4 | 7
Tongue Disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 2 | 2
Chest Pain (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 4 | 3
Gait Disturbance (General disorders) | 0 | 1 | 1 | 0
Impaired Hearing (General disorders) | 0 | 0 | 1 | 0
Influenza Like Illness (General disorders) | 0 | 0 | 1 | 0
Oedema Peripheral (General disorders) | 1 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 4
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1
Ear Infection (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 1 | 1
Herpes Zoster (Infections and infestations) | 0 | 0 | 1 | 0
Incision Site Infection (Infections and infestations) | 0 | 0 | 1 | 0
Infected Sebaceous Cyst (Infections and infestations) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Onychomycosis (Infections and infestations) | 0 | 0 | 1 | 0
Oral Herpes (Infections and infestations) | 0 | 0 | 0 | 1
Post Procedural Infection (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 1
Tooth Abscess (Infections and infestations) | 0 | 0 | 1 | 1
Tooth Infection (Infections and infestations) | 1 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 2 | 2
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 1
Anthropod Bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Confusion Postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Corneal Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 5
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Head Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Incision Site Pain (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 3
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Joint Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Meniscus Lesion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Mouth Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Post Procedural Odema (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 0 | 6 | 12
Procedural Site Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Radiation Skin Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Stress Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood Glucose Increased (Investigations) | 0 | 0 | 1 | 0
Blood Pressure Decreased (Investigations) | 0 | 0 | 0 | 1
Cardiac Murmur (Investigations) | 0 | 0 | 0 | 1
Electrocardiogram Abnormal (Investigations) | 0 | 0 | 0 | 1
Gamma-glutamyltransferase Increased (Investigations) | 0 | 0 | 0 | 1
Weight Decreased (Investigations) | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Fluid Retention (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Increased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musclar Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Osteroarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 3
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Neurilemmoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Balance Disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Cognitive Disorder (Nervous system disorders) | 0 | 0 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Drooling (Nervous system disorders) | 0 | 0 | 1 | 0
Dyskinesia (Nervous system disorders) | 2 | 2 | 6 | 5
Dystonia (Nervous system disorders) | 1 | 0 | 0 | 1
Haemorrhage Intracranial (Nervous system disorders) | 0 | 0 | 2 | 1
Headache (Nervous system disorders) | 1 | 1 | 7 | 11
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 3
Ischaemic Stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Memory Impairment (Nervous system disorders) | 0 | 0 | 3 | 3
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 3 | 0
Parkinsonism (Nervous system disorders) | 0 | 0 | 3 | 6
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0
Restless Leg Syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Sensory Disturbance (Nervous system disorders) | 0 | 0 | 0 | 1
Sleep Phase Rhythm Disturbance (Nervous system disorders) | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 2 | 1
Abnormal Dreams (Psychiatric disorders) | 1 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 2
Apathy (Psychiatric disorders) | 0 | 0 | 0 | 1
Confusional State (Psychiatric disorders) | 0 | 0 | 1 | 0
Delusions, Mixed (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 3 | 4
Disorientation (Psychiatric disorders) | 0 | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 3 | 3
Libido Increased (Psychiatric disorders) | 1 | 0 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 0 | 1
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 1
Obsessive-compulsive Disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Pathological Gambling (Psychiatric disorders) | 1 | 0 | 0 | 0
Rapid Eye Movements Sleep Abnormal (Psychiatric disorders) | 0 | 0 | 1 | 0
Social Avoidant Behavior (Psychiatric disorders) | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Micturition Urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 2 | 2
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Breast Cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Uterine Cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinitis Seasonal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dermal Cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Swelling Face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
External Fixation of Fracture (Surgical and medical procedures) | 0 | 0 | 0 | 1
Joint Surgery (Surgical and medical procedures) | 0 | 0 | 0 | 1
Tooth Extraction (Surgical and medical procedures) | 1 | 0 | 0 | 0
Varicose Vein Operation (Surgical and medical procedures) | 0 | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 1
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 2 | 0
Varicose Vein (Vascular disorders) | 0 | 0 | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No